CLINICAL TRIAL: NCT00518011
Title: A Randomized, Open Label Study Comparing the Effect of First-line Therapy With Tarceva + Gemcitabine Versus Gemcitabine Monotherapy on Treatment Response in Treatment-naïve Patients With Advanced Non-small Cell Lung Cancer
Brief Title: A Study of Tarceva (Erlotinib) and Gemcitabine in Treatment-Naive Patients With Advanced Non-Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20063
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride; Gemcitabine

ARMS (2):
- Erlotinib + Gemcitabine (Experimental): Participants received Erlotinib 150 mg/day orally as a continuous schedule with Gemcitabine 1000 (mg/m^2)/day, IV on Days 1, 8, 15 and every 4 weeks for 6 cycles.
  Interventions: Drug: Erlotinib; Drug: Gemcitabine
- Gemcitabine (Active Comparator): Participants received Gemcitabine 1000 (mg/m^2)/day, IV on Days 1, 8, 15 and every 4 weeks for 6 cycles.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Erlotinib — 150 mg po daily
  Arms: Erlotinib + Gemcitabine
Drug: Gemcitabine — As prescribed

SUMMARY:
This 2 arm study will assess the efficacy and safety of Tarceva plus gemcitabine, compared with gemcitabine alone, in the treatment of chemotherapy-naive patients with advanced non-small cell lung cancer. Patients will be randomized to receive either Tarceva 150mg po daily plus gemcitabine on days 1, 8, 15 and every 4 weeks subsequently, or with gemcitabine monotherapy. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* non-small cell lung cancer, stage IIIb (with effusion) or stage IV with measurable disease ;
* ECOG PS 2;
* adequate organ function.

Exclusion Criteria:

* prior chemotherapy or systemic anti-tumor therapy;
* hypersensitivity to erlotinib;
* any condition contraindicating the use of the study medication and/or impairing the interpretation of results and/or leading to treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Australia (13):
  - Auchenflower
  - Chermside
  - Footscray
  - Greenslopes
  - Lismore
  - Melbourne
  - Parkville
  - Randwick
  - Richmond
  - St Leonards
  - Sydney
  - Wodonga
  - Wollongong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 chemo-naïve participants with Non-Small Cell Lung Cancer (NSCLC) Stage IIIB with pleural effusion or stage IV and a Eastern Cooperative Oncology Group performance status 2 (PS 2) were recruited. The study was conducted from 24 August 2007 to 14 February 2009 at 14 Centers in Australia.
Pre-assignment Details: Total 17 participants were enrolled; however the data was available for 16 participants. One participant in the gemcitabine arm withdrew consent before receiving treatment.
Groups:
- Gemcitabine: Participants received Gemcitabine 1000 milligram per meter square (mg/m^2)/day, intravenously (IV) on Days 1, 8, 15 and every 4 weeks for 6 cycles
Period: Overall Study
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Started | 9 | 8
Completed | 0 | 0
Not Completed | 9 | 8
Not completed — Death | 1 | 1
Not completed — Adverse Event | 2 | 3
Not completed — Disease Progression | 2 | 2
Not completed — Other Reasons | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics were analyzed using the intention-to-treat (ITT) population. ITT included all randomized participants.
  years | 71.6 (12.94) | 76.8 (4.17) | 74.0 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival was defined as the interval between the day of randomization and the date of the first documentation of disease progression or date of death (from any cause), whichever occurs first.
Time Frame: Up to 2 years
Population: Per protocol (PP) population included all randomized participants who received at least one dose of study medication and had at least one post baseline tumor assessment or record of death.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Number analyzed (Participants) | 8 | 7
Week | 23.3 [7.1 to 24.9] | 24.4 [6.9 to NA] — Not evaluable due to insufficient follow-up time and / or insufficient number of events.
Statistical Analysis 1: Comparison: Gemcitabine vs Erlotinib + Gemcitabine; Test type: Superiority or Other; p = 0.3644, Log Rank; Hazard Ratio (HR) = 1.842, 95% CI 2-sided [0.483 to 7.027]

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants who have any evidence of confirmed objective of complete response (CR) + partial response (PR), as assessed by the Response Evaluation Criteria In Solid Tumors (RECIST version 1.0) criteria. As per the RECIST Version 1.0 CR is defined as disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of the LD.
Time Frame: Up to 2 years
Population: PP population included all randomized participants who received at least one dose of study medication and had at least one post baseline tumor assessment or record of death.
Measure: Number; unit: Percentage of participants
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Number analyzed (Participants) | 8 | 7
Percentage of participants | 0 | 28.6

3. Secondary Outcome: Disease Control Rate
Description: Disease control rate was defined as the percentage of participants who have any evidence of confirmed objective CR or PR or Stable disease (SD) (where SD was maintained for 8 weeks), as assessed by the RECIST version 1.0 criteria. As per the RECIST Version 1.0 CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum of the LD. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum of the LD since the treatment started. PD is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum of the LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Number analyzed (Participants) | 8 | 7
Percentage of participants | 50 | 85.7

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the interval between the date of CR or PR was first recorded to the date on which progressive disease was first noted or date of death.
Time Frame: Up to 2 years
Population: PP population included all randomized participants received at least one dose of study medication and had at least one post baseline tumor assessment or record of death. Participants available at the time of evaluation of duration of response were included in the analysis.
Measure: Mean (Standard Deviation); unit: Week
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Number analyzed (Participants) | 0 | 2
Week |  | 16.3 (NA) — Not evaluable due to insufficient follow-up time and / or insufficient number of events.

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval between the date of randomization to the date of death from any cause.
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Number analyzed (Participants) | 8 | 7
Week | 21.1 [7.6 to NA] — Not evaluable due to insufficient follow-up time and / or insufficient number of events. | 39.0 [6.9 to NA] — Not evaluable due to insufficient follow-up time and / or insufficient number of events.
Statistical Analysis 1: Comparison: Gemcitabine vs Erlotinib + Gemcitabine; Test type: Superiority or Other; p = 0.7165, Log Rank; Hazard Ratio (HR) = 1.278, 95% CI 2-sided [0.339 to 4.824]

6. Secondary Outcome: Mean Change in Pulse Rate From Baseline
Description: Mean change in pulse rate from Baseline for each cycle calculated as Day 1 of each cycle value minus Baseline value
Time Frame: Baseline (Day -14 to Day 0), Cycle 1 (Days 1, 8, 15 and 22), Cycle 2 (Days 1, 8, 15 and 22), Cycle 3 (Days 1, 8, and 15), Cycle 4 (Days 1, 8, and 15), Cycle 5 (Days 1, 8, and 15), Cycle 6 (Days 1, 8, and 15)
Population: Safety population included all participants who received at least one dose or infusion of study treatment and had a safety assessment performed at baseline.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Number analyzed (Participants) | 8 | 8
beats per minute
  Cycle 1 (n=8, 8) | 2.37 (14.31) | 3.00 (5.58)
  Cycle 2 (n=7, 6) | 3.00 (12.19) | -3.00 (12.96)
  Cycle 3 (n=4, 5) | 2.75 (13.14) | -1.80 (7.08)
  Cycle 4 (n=1, 5) | 18.00 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | 1.80 (15.33)
  Cycle 5 (n=1, 3) | -6.00 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | -9.00 (18.52)
  Cycle 6 (n= 1, 2) | 4.00 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | 6.00 (0.00)

7. Secondary Outcome: Mean Change in Blood Pressure From Baseline
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were recorded as vital parameters in this study. Mean change in SBP and DBP from Baseline for each cycle calculated as Day 1 of each cycle value minus baseline value.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Number analyzed (Participants) | 8 | 8
mm Hg
  SBP at Cycle 1 (n=8, 8) | 3.00 (6.34) | -0.87 (9.40)
  DBP at Cycle 1 (n=8, 8) | -6.87 (9.41) | -5.37 (12.21)
  SBP at Cycle 2 (n=7, 6) | -4.85 (8.33) | -17.83 (9.90)
  DBP at Cycle 2 (n=7, 6) | -10.71 (9.44) | -9.50 (11.81)
  SBP at Cycle 3 (n=4, 5) | -9.00 (8.67) | -17.20 (19.14)
  DBP at Cycle 3 (n=4, 5) | -8.25 (11.89) | -9.20 (15.64)
  SBP at Cycle 4 (n=1, 5) | -18.00 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | -10.20 (16.52)
  DBP at Cycle 4 (n=1, 5) | -4.00 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | -1.60 (14.32)
  SBP at Cycle 5 (n=1, 3) | 28.00 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | -1.66 (12.34)
  DBP at Cycle 5 (n=1, 3) | 12.00 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | 0.66 (2.51)
  SBP at Cycle 6 (n=1, 2) | 10.00 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | 5.00 (0.00)
  DBP at Cycle 6 (n=1, 2) | 5.00 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | -0.50 (2.12)

8. Secondary Outcome: Mean Change in Body Temperature From Baseline
Description: Mean change in body temperature from Baseline for each cycle calculated as Day 1 of each cycle value minus baseline value.
Time Frame: as for outcome 6
Population: Safety population included all participants who received at least one dose/infusion and had at least one safety assessment performed at baseline.
Measure: Mean (Standard Deviation); unit: Fahrenheit
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Number analyzed (Participants) | 8 | 8
Fahrenheit
  Cycle 1 (n=8, 8) | -0.02 (0.73) | -0.012 (0.11)
  Cycle 2 (n=7, 6) | 0.14 (0.82) | -0.30 (0.40)
  Cycle 3 (n=4, 5) | -0.07 (0.68) | -0.32 (0.37)
  Cycle 4 (n=1, 5) | -0.60 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | -0.24 (0.46)
  Cycle 5 (n=1, 3) | -0.70 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | -0.46 (0.25)
  Cycle 6 (n=1, 2) | -0.20 (NA) — Standard Deviation was not calculated as only single participant was present for this group. | -0.20 (0.98)

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse event is defined as any untoward medical occurrence in a patient administered a pharmaceutical product and includes any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Groups:
- Gemcitabine: Participants received Gemcitabine (1000 mg/m^2/day), IV on Days 1, 8, 15 of each 4 week cycle for 6 cycles
Arm/Group | Gemcitabine | Erlotinib + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 5/8 | 6/8
Other Adverse Events (participants affected / at risk) | 7/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (N=8) | Erlotinib + Gemcitabine (N=8)
Pneumonia (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Recall phenomenon (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1 — General disorders and administration site conditions
Oedema peripheral (General disorders) | 0 | 1 — General disorders and administration site conditions
Pain (General disorders) | 0 | 1 — General disorders and administration site conditions
Pyrexia (General disorders) | 0 | 1 — General disorders and administration site conditions
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (N=8) | Erlotinib + Gemcitabine (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Nausea (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 4 | 4 — General disorders and administration site conditions
Oedema peripheral (General disorders) | 1 | 2 — General disorders and administration site conditions
Chills (General disorders) | 1 | 0 — General disorders and administration site conditions
Feeling cold (General disorders) | 0 | 1 — General disorders and administration site conditions
Influenza like illness (General disorders) | 1 | 0 — General disorders and administration site conditions
Malaise (General disorders) | 1 | 0 — General disorders and administration site conditions
Mucosal inflammation (General disorders) | 0 | 1 — General disorders and administration site conditions
Pain (General disorders) | 0 | 1 — General disorders and administration site conditions
Pyrexia (General disorders) | 0 | 1 — General disorders and administration site conditions
Haemoglobin decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose fluctuation (Investigations) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 3
Dysphasia (Nervous system disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 1
Penile swelling (Reproductive system and breast disorders) | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1
Cerebral hygroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.